CLINICAL TRIAL: NCT01459341
Title: Comparison of Near Infrared Spectroscopy (NIRS) and Transcutaneous Oxygen Pressure (TCPO2) Measurements in Critical Limb Ischemia (CLI) Patients After Invasive Treatment (Endovascular or Surgery)
Brief Title: Near Infrared Spectroscopy and Transcutaneous Oxygen Pressure in Critical Limb Ischemia Before and After Treatment
Acronym: NIRS
Status: Completed | Type: Observational
Sponsor: Carmel Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: CMC-11-0017 CTIL; NIRS-001-Carmel (Other: Carmel Medical Center)
Record Dates: First submitted 2011-10-18; First posted 2011-10-25 (Estimated); Last update posted 2012-12-06 (Estimated); Status verified 2012-12

CONDITIONS: Peripheral Vascular Disease; Critical Limb Ischemia
Keywords: CLI Critical limb ischemia; PVD peripheral vascular disease; NIRS near infrared spectroscopy; TCPO2 - transcutaneous oxygen pressure
MeSH Terms: conditions — Peripheral Vascular Diseases; Chronic Limb-Threatening Ischemia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Comparison of two non-invasive methods for measuring tissue oxygenation. One is Transcutaneous Oxygen Pressure (TCPO2) and the other is the new method of Near Infrared Spectroscopy (NIRS) - near infrared spectroscopy in patients with critical limb ischemia (CLI) undergoing invasive treatment (surgical or endovascular).

DETAILED DESCRIPTION:
Comparison of two non-invasive methods for measuring tissue oxygenation. One is TCPO2 and the other is the new method of NIRS - near infrared spectroscopy in patients with critical limb ischemia (CLI) undergoing invasive treatment (surgical or endovascular).

The NIRS probe has been used to measure tissue oxygenation in the cerebral circulation up to now. While TCPO2 is the established method for measuring tissue oxygenation in patients with CLI to evaluate the potential for wound healing.

ELIGIBILITY:
Inclusion Criteria:

* 10 patients admitted to the vascular surgical department and undergoing invasive treatment (surgical or endovascular)

Exclusion Criteria:

* pregnancy allergy to iod advanced renal failure CCT<50 active peptic ulcer recent bleeding

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 10 patients admitted to the vascular surgical department and undergoing invasive treatment (surgical or endovacular)
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2011-07; Primary Completion 2012-09 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
tissue oxygenation | the outcome will be assessed during the hospital stay up to a week

CONTACTS AND LOCATIONS:
Overall Officials: Dallit Mannheim, MD, Principal Investigator — Carmel Medical Center
Locations (1):
- department of vascular surgery, Carmel medical center, Haifa, Israel

REFERENCES:
- [Result] Murkin JM, Arango M. Near-infrared spectroscopy as an index of brain and tissue oxygenation. Br J Anaesth. 2009 Dec;103 Suppl 1:i3-13. doi: 10.1093/bja/aep299. PMID 20007987